CLINICAL TRIAL: NCT06561152
Title: Tagraxofusp and Low-Intensity Chemotherapy for the Treatment of CD123-Positive Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Tagraxofusp and Low-Intensity Chemotherapy for CD123-Positive Relapsed or Refractory AML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Gabriel Mannis, Associate Professor of Medicine (Hematology), Stanford University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-76512
Record Dates: First submitted 2024-08-16; First posted 2024-08-19 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Refractory Acute Myeloid Leukemia; Relapsed Acute Myeloid Leukemia
Keywords: tagraxofusp; cladribine; cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tagraxofusp; Cladribine; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose level 1 (DL1) (Experimental): DL1 will consist of cladribine 5mg/m2 IV once daily on days 1-3, cytarabine 20mg/m2 IV daily days 1-5, and tagraxofusp 12 mcg/kg IV daily days 4-6. If a DLT is encountered in the first 2 participants, 3 more will be enrolled at the same dose.
  Interventions: Drug: Tagraxofusp; Drug: Cladribine (CLAD); Drug: Cytarabine
- Dose level 2 (DL2) (Experimental): DL2 will consist of cladribine 5mg/m2 IV once daily on days 1-4, cytarabine 20mg/m2 IV daily days 1-7, and tagraxofusp 12 mcg/kg IV daily days 4-6. If a DLT is encountered in the first 2 participants, 3 more will be enrolled at the same dose.
  Interventions: Drug: Tagraxofusp; Drug: Cladribine (CLAD); Drug: Cytarabine
- Dose level 3 (DL3) (Experimental): DL3 will consist of cladribine 5mg/m2 IV once daily on days 1-5, cytarabine 20mg/m2 IV daily days 1-10, and tagraxofusp 12 mcg/kg IV daily days 4-6. If a DLT is encountered in the first 2 participants, 3 more will be enrolled at the same dose.
  Interventions: Drug: Tagraxofusp; Drug: Cladribine (CLAD); Drug: Cytarabine
- Dose Level -1 (DL-1) (Experimental): DL -1 will consist of cladribine 5mg/m2 IV once daily on days 1-2, cytarabine 20mg/m2 IV daily days 1-4, and tagraxofusp 12mcg/kg IV daily days 4-6.
  Interventions: Drug: Tagraxofusp; Drug: Cladribine (CLAD); Drug: Cytarabine

INTERVENTIONS:
Drug: Tagraxofusp — Tagraxofusp is administered by intravenous infusion (IV) over 15 minutes for 3 consecutive days of a 28-day cycle. (days 4-6)
Drug: Cladribine (CLAD) — Cladribine 5mg/m2 IV once daily on days 1-3 (DL1) Cladribine 5mg/m2 IV once daily on days 1-4 (DL2) Cladribine 5mg/m2 IV once daily on days 1-5 (DL3)
Drug: Cytarabine — Cytarabine 20mg/m2 IV daily days 1-5 (DL1) Cytarabine 20mg/m2 IV daily days 1-7(DL2) cytarabine 20mg/m2 IV daily days 1-10 (DL3)

SUMMARY:
To determine the efficacy of the combination of tagraxofusp, cladribine, and cytarabine.

ELIGIBILITY:
Inclusion Criteria

* Documented diagnosis of relapsed or refractory acute myeloid leukemia (AML) according to World Health Organization (WHO) 2022 criteria
* Expression of CD123 by either flow cytometry or immunohistochemical staining with no minimum threshold for positivity
* Must have received initial therapy with venetoclax in combination with a hypomethylating agent (either azacitidine or decitabine) with no subsequent therapy unless mutations in the IDH or FLT3 genes.

If mutations in the IDH or FLT3 genes, treatment with IDH or FLT3 inhibitors after initial failure of venetoclax plus HMA is allowed, but not required.

* Age ≥ 18 years of age
* ECOG ≤ 2
* Albumin ≥ 3.2 g/dL at time of screening (note that albumin supplementation is not permitted to enable eligibility)
* Left ventricular ejection fraction ≥ 50%
* No clinically significant abnormalities on 12-lead electrocardiogram (ECG) including: complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250ms, or QTcF (Friderica's method) >450ms in 3 successive measurements
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Females of reproductive potential need to either commit to true abstinence from heterosexual contact or agree to use, and be able to comply with highly effective contraception without interruption prior to starting treatment, during the study therapy, and for 30 days after last dose of study therapy
* For males of reproductive potential: agreement to use of condoms
* Adequate hepatic/renal function defined as:

Hepatic function: total bilirubin ≤ 1.5 x ULN (unless attributable to Gilbert's disease or leukemic involvement) AND AST or ALT ≤ 3 x ULN

Renal function: creatinine clearance > 30 mL/minute, calculated by Cockcroft Gault formula

* Women of childbearing potential must have a negative urine or serum pregnancy test
* Ability to understand and the willingness to provide written informed consent.

Exclusion Criteria:

* Prior therapy apart from Venetoclax in combination with a hypomethylating agent, or Venetoclax in combination with a hypomethylating agent followed by monotherapy with IDH or FLT3 inhibitors
* Patients who received systemic anti-cancer therapy <14 days prior to their first day of study drug administration.
* Patients who received systemic anti-cancer therapy <14 days prior to their first day of study drug administration. Concurrent hydroxyurea will be allowed. Hydroxyurea use will be allowed only during the first cycle if needed for disease control.
* Significant cardiac disease (any NYHA Class 3 or 4 CHF, uncontrolled angina, history of MI, unstable angina or stroke within 6 months prior to study entry, uncontrolled hypertension, or clinically significant arrhythmias not controlled by medication)
* Any uncontrolled bacterial, fungal, viral or other infection.
* Known HIV+ or active hepatitis B or C infection, defined as positive viral load for HBV or HCV or a positive surface antigen (HBsAg) test for hepatitis B.
* The patient has persistent clinically significant toxicities Grade >/= 2 from previous therapies not readily controlled by supportive measures (excluding alopecia, nausea, and fatigue).
* The patient has an active malignancy and/or cancer history that may confound the assessment of the study endpoints. Patients with a past cancer history (within 2 years of study entry) with substantial potential for recurrence and/or ongoing active malignancy must be discussed with study team before study entry. Patients with the following neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ, cervical intraepithelial neoplasia, organ-confined prostate cancer with no evidence of progressive disease.
* The patient has uncontrolled, clinically significant pulmonary disease (e.g. chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the Investigator would put the patient at significant risk for pulmonary complications during the study.
* The patient has known active or suspected CNS disease. If suspected, CNS disease should be ruled out with relevant imaging and/or examination of cerebrospinal fluid.
* The patient is receiving immunosuppressive therapy - with the exception of low-dose prednisone (</= 10 mg/day).
* Received allogenic stem cell transplant prior to the treatment.
* The patient has an uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 dose | up 2 years
  Determination of the recommended Phase 2 dose based on the safety of tagraxofusp in combination with cladribine and low-dose cyatarabine, as determined by DLT evaluation.

SECONDARY OUTCOMES:
Overall response rate (ORR) | up 2 years
  ORR will be determined by the proportion of study subjects achieving Complete Remission (CR), Complete remission with incomplete hematologic recovery (CRi), Complete remission with partial hematologic recovery (CRh), Morphological leukemia-free state (MLFS), or (Partial Response (PR), as defined by the ELN 2022 AML response criteria.
Complete response | up 2 years
  Complete Response will be determined by the proportion of study subjects achieving CR, as defined by the ELN 2022 AML Response Criteria.
Composite complete response (CR+CRi +CRh) | up 2 years
  Composite complete response will be determined by the proportion of study subjects achieving CR, CRi, or CRh, as defined by the ELN 2022 AML Response Criteria.
Rate of Minimal Residual Disease (MRD) negativity in responders | up 2 years
  Rate of MRD negativity in responders, as measured by multi-parameter flow cytometry.
Duration of overall survival | up 2 years
  Overall survival (OS) will be measured as the date of enrollment in the study to the date of death from any cause.
Incidence of drug-related adverse events | up 2 years
  The Incidence of Drug-Related Adverse Events is a safety endpoint used to evaluate the frequency and severity of adverse events (AEs) that are attributed to the study drug All grades of adverse events determined to be treatment-related will be summarized descriptively.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States